CLINICAL TRIAL: NCT03976076
Title: A Phase 2 Study to Assess the Safety, Tolerability, Exploratory Efficacy, and Pharmacokinetics of Orally Administered JBPOS0101 for Refractory Infantile Spasms Patients
Brief Title: A Study of Orally Administered JBPOS0101 in Refractory Infantile Spasms Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with patient recruitment due to COVID-19
Sponsor: Bio-Pharm Solutions Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-0101-WS01
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Refractory Infantile Spasms
Keywords: JBPOS0101; Infantile Spasms; Electroencephalogram
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Intervention Model Description: Patients received the investigational product at a dose of 6 milligram per kg orally twice daily; once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on the day of Visit 3, the dose was escalated and patients received the investigational product at a dose of 9 mg/kg orally twice daily. Starting on Day 15, the dose was escalated again and patients received the investigational product at a dose of 15 mg/kg orally twice daily until the end of Treatment Period 1 (Day 28).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JBPOS0101 (investigational product) (Experimental): During Treatment Period 1, the IP was administered at 6 mg/kg, per oral (PO), twice a day (BID), once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the Investigational Product (JBPOS0101) (IP) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing.
  Interventions: Drug: JBPOS0101

INTERVENTIONS:
Drug: JBPOS0101 — JBPOS0101 (investigational product)

SUMMARY:
A Phase 2 Study to Assess the Safety, Tolerability, Exploratory Efficacy, and pharmacokinetics of Orally Administered JBPOS0101 for Refractory Infantile Spasms Patients.

DETAILED DESCRIPTION:
This open label, multicenter study allowed JBPOS0101 (investigational product) to be given as either add-on therapy or monotherapy for patients with refractory infantile spasms. The design and choice of study population of this Phase 2 clinical study was based on the need to provide initial safety, tolerability, pharmacokinetics (PK), and efficacy outcomes of the investigational product for future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 6 months through 36 months of age at the time of informed consent
* Had clinical diagnosis of Infantile spasms (IS), confirmed by video-electroencephalogram (EEG) analysis, and hypsarrhythmia on EEG at screening according to the Burden of Amplitudes and Epileptiform Discharges (BASED) scale score.
* As assessed by the investigator had no or partial response to at least 2 out of the 3 therapies of adrenocorticotrophic hormone (ACTH), vigabatrin, and glucocorticoids (i.e. prednisolone), or had no or partial response to at least 1 out of the 3 therapies of ACTH, vigabatrin, and glucocorticoids and was contraindicated to and/or refused by the patient's legal representative(s) for treatment with one or both other 2 therapies.
* Patient had general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on physical and neurological examinations, medical history, normal renal function and electrocardiogram (ECG), and clinical laboratory values completed during the Screening Period visit (Visit 1).
* Parent(s)/caregiver(s) were willing and able to comply with the study procedures and visit schedules in the opinion of the investigator.
* Parent(s)/caregiver(s) fully comprehend and sign the ICF in accordance with applicable laws, regulations, and local requirements, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator.

Exclusion Criteria:

* Patient considered by the investigator, for any reason (including, but not limited to, the risks described as precautions and warnings in the current version of the investigator's brochure for investigational product) to be an unsuitable candidate to receive the investigational product.
* Patient had known or suspected allergy to the investigational product or apple juice.
* Patient had clinically significant renal impairment, defined as creatinine >1.5 mg/dL or blood urea nitrogen >2 × upper limit of normal (ULN);
* Clinically significant liver dysfunction, defined as total bilirubin ≥2 × ULN, or aspartate aminotransferase or alanine aminotransferase ≥3 × ULN;
* Patient had clinically significant abnormal laboratory values; the investigator may deem the patient eligible if he/she judges the laboratory values to be not clinically significant.
* Patient had an ongoing or known history of human immunodeficiency virus infection, or chronic hepatitis B or C.
* Patient had a clinically significant abnormality on ECG that, in the opinion of the investigator, increases the safety risks of participating in the study.
* Patient had a neurodegenerative disorder as the underlying cause of IS.
* Patient had a known history of aspiration pneumonia within the past year.
* Patient had previously participated in another clinical study of the investigational product or received any investigational drug or device or investigational therapy within 30 days of study entry.
* Patient had received therapy with felbamate, cannabinoids, ketogenic diet or vagus nerve stimulation within 14 days of screening.
* Patient had received therapy with a medication known to be a CYP3A4 substrate and whose PK had been shown to be impacted in the presence of a CYP3A4 inhibitor within 14 days of screening.
* Patient had not remained at stables doses of all drugs used for treating epileptic seizures for at least 14 days prior to screening (except for rescue medications used for acute treatment of breakthrough seizures which were not known to be CYP3A4 substrates and whose PK had not been shown to be impacted in the presence of a CYP3A4 inhibitor.
* Patient had a lethal or potentially lethal condition other than infantile spasms, with a significant risk of death before 18 months of age such as non-ketotic hyperglycinemia.
* Patient had a body weight below 5 kg.
* Patient had an underlying metabolic disease associated with glucose intolerance (e.g., glucose transporter deficiencies).

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Kim, Study Director — Bio-Pharm Solutions
Locations (23):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital LA, Los Angeles, California
  - UCLA - David Geffen School of Medicine, Los Angeles, California
  - UCSF Epilepsy Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Neurology, PA, Winter Park, Florida
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Multicare Institute for Research and Innovation, Tacoma, Washington
- South Korea (6):
  - Pusan National University Yangsan Hospital, Pusan, Gyeongsangnam-do
  - Kyungpook National University Chilgok Hospital (KNUH), Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible patients (met all the inclusion and none of the exclusion criteria) whose legal representative (parent[s]/caregiver[s]) provided a written informed consent were enrolled in the study and entered the treatment period on Day 1. Patients were recruited from 15 April 2020 to 10 Dec 2021 for this study.
Pre-assignment Details: An overnight video-EEG was completed within the Screening Period (Days -28 to -6) and repeated at Day 28 (Visit 5 [± 2 days]), following Treatment Period 1 for assessment of spasms and hypsarrhythmia. Sixteen participants were actually enrolled, of whom 12 participants were treated. Four patients were screen failures; (2 patients failed to meet the inclusion/exclusion criteria and 2 patients were screen failed due to the other reasons).
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6mg/kg, per oral (PO), twice a day (BID), once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the Investigational Product (JBPOS0101) (IP) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was100 mg, white to off-white powder for reconstitution into an oral solution.
Period: Overall Study
Arm/Group | JBPOS0101 (Investigational Product)
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6mg/kg, PO, BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the IP (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.93 (8.373)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any event that did not present before exposure to the investigational product (IP) or any event already present that worsened in either intensity or frequency after exposure to the IP.
Time Frame: Day 1 to Day 56
Population: Safety Population: Included all patients who were treated with at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, PO, twice a BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the IP (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 12
Participants | 12

2. Secondary Outcome: JBPOS0101 Plasma Concentration 0.5 - 1.5 Hours Post Morning Dose, Day 1
Description: Pharmacokinetics: JBPOS0101 plasma concentration 0.5 - 1.5 hours post morning dose on Day 1
Time Frame: 0.5 to1.5 hours post morning (AM) dose on Day 1
Population: PK population: The PK population included all patients, without any major protocol deviation affecting the secondary endpoint analysis, who were treated with at least one dose of the IP and had at least one measurable PK concentration.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, PO, BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the IP (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 12
Nanograms per milliliter (ng/mL) | 6150.0 (1845.45)

3. Secondary Outcome: JBPOS0101 Plasma Concentration 4-6 Hours Post Morning Dose, Day 1
Description: Pharmacokinetics: JBPOS0101 plasma concentration 4 - 6 hours post morning dose on Day 1
Time Frame: 4 to 6 hours post morning (AM) dose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, per oral, BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the IP (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was 100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 12
ng/mL | 5854.2 (904.85)

4. Secondary Outcome: JBPOS0101 Plasma Concentration 8 Hours Post Morning Dose and Pre-PM Dose, Day 1
Description: Pharmacokinetics: JBPOS0101 plasma concentration 8 hours post morning dose and pre-PM dose on Day 1.
Time Frame: 8 hours post morning (AM) dose and pre-PM dose on Day 1
Population: PK population: The PK population included all patients, without any major protocol deviation affecting the secondary endpoint analysis, who were treated with at least one dose of the IP and had at least one measurable PK concentration. Here N=12 is the overall number of participants. n= 11 signifies number of participants with available data for specified time.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, per oral, BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the IP (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP is 100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 11
ng/mL | 4172.7 (765.13)

5. Secondary Outcome: JBPOS0101 Plasma Concentration 0.5 -1.5 Hours Post Morning Dose, Day 21
Description: Pharmacokinetics: JBPOS0101 plasma concentration 0.5 - 1.5 hours post morning dose on Day 21
Time Frame: 0.5 to1.5 hours post morning (AM) dose on Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 11
ng/mL | 22945.5 (3599.27)

6. Secondary Outcome: JBPOS0101 Plasma Concentration 4 - 6 Hours Post Morning Dose, Day 21
Description: Pharmacokinetics: JBPOS0101 plasma concentration 4 - 6 hours post morning dose on Day 21
Time Frame: 4 to 6 hours post morning (AM) dose on Day 21
Population: PK population: PK Population: The PK population included all patients, without any major protocol deviation affecting the secondary endpoint analysis, who were treated with at least one dose of the IP and had at least one measurable PK concentration.
  Here N=12 is the overall number of participants. n= 10 signifies number of participants with available data for specified time.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, PO, BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the IP (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was 100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 10
ng/mL | 18070.0 (4184.11)

7. Secondary Outcome: JBPOS0101 Plasma Concentration 8 Hours Post Morning Dose and Pre-PM Dose, Day 21
Description: Pharmacokinetics: JBPOS0101 plasma concentration 8 hours post morning dose and pre-PM dose on Day 21.
Time Frame: 8 hours post morning (AM) dose and pre-PM dose on Day 21
Population: PK population: PK Population: The PK population included all patients, without any major protocol deviation affecting the secondary endpoint analysis, who were treated with at least one dose of the IP and had at least one measurable PK concentration.
  Here N=12 is the overall number of participants. n= 9 signifies number of participants with available data for specified time.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, per oral (PO), twice a day (BID), once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the Investigational Product (JBPOS0101) (IP) at a dose of 9 mg/kg orally BID. Starting on Day 15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 9
ng/mL | 12921.1 (3220.22)

8. Secondary Outcome: JBPOS0101 Urine Concentration at Day 1
Description: Pharmacokinetics: JBPOS0101 urine concentration on Day 1. Urine samples were collected following the morning dose.
Time Frame: Day 1
Population: PK population: The PK population included all patients, without any major protocol deviation affecting the secondary endpoint analysis, who were treated with at least one dose of the IP and had at least one measurable PK concentration. Here N=12 is the overall number of participants. n= 10 signifies number of participants with available data for specified time.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 10
ng/mL | 3410.0 (1152.50)

9. Secondary Outcome: JBPOS0101 Urine Concentrations at Day 21
Description: Pharmacokinetics: JBPOS0101 urine concentration on Day 21. Urine samples were collected following the morning dose.
Time Frame: Day 21
Population: PK population: The PK population included all patients, without any major protocol deviation affecting the secondary endpoint analysis, who were treated with at least one dose of the IP and had at least one measurable PK concentration. Here N=12 is the overall number of participants. n= 9 signifies number of participants with available data for specified time.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JBPOS0101 (Investigational Product)
Number analyzed (Participants) | 9
ng/mL | 14360.0 (6986.77)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 56.
Description: Adverse event analyses were conducted on the safety population. A treatment-emergent adverse event (TEAE) was defined as any AE that began or worsened following the start of dosing of Treatment Period 1, Day 1 to Follow-Up.
  NOTE:
  Seizure (SAE) and aspiration pneumonia (SAE) were not related to IP. The investigator noted for the TEAE "Electrocardiogram QT prolonged" that the patient was distressed and crying to the point of hyperventilation.
Groups:
- JBPOS0101 (Investigational Product): JBPOS0101: JBPOS0101 (investigational product)
  During Treatment Period 1, the IP was administered at 6 mg/kg, PO, BID, once in the morning and 12 hours following the morning dose during the first 7 days of Treatment Period 1. Starting from the PM dose on Visit 3, the dose was escalated and patients received the Investigational Product (JBPOS0101) at a dose of 9 mg/kg orally BID. Starting on Day15, the dose was escalated again and patients received the IP at a dose of 15 mg/kg orally BID until the end of Treatment Period 1 (Day 28). Each dose of the IP was administered after at least a 2-hour fast. Food was given 2 hours after dosing. IP was 100 mg, white to off-white powder for reconstitution into an oral solution.
Arm/Group | JBPOS0101 (Investigational Product)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JBPOS0101 (Investigational Product) (N=12)
Liver function test increased (Investigations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JBPOS0101 (Investigational Product) (N=12)
Somnolence (Nervous system disorders) | 3 (3)
Sedation (Nervous system disorders) | 2 (4)
Liver function test increased (Investigations) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Sedation complication (Injury, poisoning and procedural complications) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Drooling (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Pyrexia (General disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2)
Otitis media acute (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations reported for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03976076/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03976076/SAP_001.pdf